CLINICAL TRIAL: NCT06222190
Title: Online-adaptive Radiotherapy in Lung Cancer
Brief Title: Lung_Cancer_adaptive - Ethos
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: UME-ID-11766
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: online-adaptive radiotherapy — A conebeam CT is taken to determine the current tumour extent and the deformations occurring in comparison to the dose distribution to be applied. Normal tissues heart, lung and tracheal tree are automatically contoured by the Ethos therapy system in that cone-beam CT. A specialist physician and a physicist are present during this process. These organ contours are used to determine the extent of the current target volume and the adaptive radiotherapy plan is adjusted to the new target volume. If the current tumour extent is not sufficiently covered by the initial radiotherapy plan planned for the series with its planned tolerances, or if the surrounding normal tissue is exposed to too much radiation, then the online adaptive radiotherapy plan for the current treatment is selected by the specialist. Otherwise, the initial radiotherapy plan is used for IGRT.
  Other Names: ETHOS therapy system (Varian Medical Systems)

SUMMARY:
In patients with lung carcinoma who receive radiotherapy preoperatively or alternatively curative, high-dose radiotherapy instead of surgery, there are also deformations of the thorax from fraction to fraction.

Currently, ART for lung carcinomas is carried out as part of patient care in the radiotherapy clinic. Patients are irradiated during repeated breath-holding manoeuvres in deep inspiration. The breath-holding manoeuvre is practised several times before the daily irradiation. An optical surface detection device is available for this purpose, which is used to compare the body surface in the patient's thorax area on the treatment table with the target surface to be achieved during radiotherapy planning, which took place days before the current fraction. If the target surface is reproducibly achieved, a conebeam CT is taken to determine the current tumour extent and the deformations occurring in comparison to the dose distribution to be applied. For this purpose, the normal tissues heart, lung and tracheal tree are automatically contoured by the Ethos therapy system in the cone-beam CT. A specialist physician and a physicist are present at the Ethos device during this process. These organ contours are used to determine the extent of the current target volume and the adaptive radiotherapy plan is adjusted to the new target volume. If the current tumour extent is not sufficiently covered by the initial radiotherapy plan planned for the series with its planned tolerances, or if the surrounding normal tissue is exposed to too much radiation, then the online adaptive radiotherapy plan for the current treatment is selected by the specialist. Otherwise, the initial radiotherapy plan is used by the planning CT as for IGRT.

The aim of this study is to treat patients in ART readiness on the Ethos therapy device over 10 radiotherapy fractions. The dose distribution is always compared with the adaptive and the initial series plan on the anatomy of the day by the specialist and medical physics expert. The ART plan is applied when dosimetric advantages are present. The aim of this study is to prospectively analyse in how many patients safety margins around the clinical target volume can be reduced with ART compared to IGRT. The percentage of patients who benefit from ART will be determined prospectively. The criterion for a relevant benefit from ART is the effective uniform dose (EUD) in the target volume with the accumulated dose distribution across the first 7 fractions. If the EUD is below 95% of the target dose with IGRT and above 95% of the target dose with ART, then an advantage is determined with ART. Patients with a benefit from ART receive ART for the further fractions of the series, while the others continue to be treated with IGRT.

DETAILED DESCRIPTION:
With online-adaptive radiotherapy (ART), the radiotherapy plan can be adapted to the anatomical changes before each radiotherapy fraction. The basis for adaptation is a cone-beam CT with the patient on the treatment table at the start of each radiotherapy fraction. Adaptive radiotherapy is a further development of image-guided radiotherapy (IGRT), which is now the basic standard in radiotherapy. Here, a cone beam CT is also performed at the start of each fraction, but this is only used to position the patient in relation to the radiation field arrangement of the initial radiation plan approved for the series, so that predefined landmarks match the target position in the planning CT as closely as possible. However, the radiotherapy plan itself cannot be adapted to deformations in the body during IGRT, e.g. due to different bowel and bladder fillings. IGRT is currently carried out on all linear accelerators at the radiotherapy clinic. For online adaptive radiotherapy (ART), which allows the radiotherapy plan to be adapted to the anatomical deformities of the day online on the treatment table, the ETHOS® radiotherapy system from Varian-Siemens has been available at the radiotherapy clinic for a year as a medical device with handling authorisation from the district government. This therapy device enables on-line adaptive plan adjustment within 10-20 minutes.

In patients with lung carcinoma who receive radiotherapy preoperatively to reduce the size of the tumour before surgery or alternatively curative, high-dose radiotherapy instead of surgery, there are also deformations of the thorax from fraction to fraction. For example, the depth of breathing during deep inspiration radiotherapy can change depending on the shape of the day. Ventilation disturbances caused by the tumour may increase or decrease, pleural effusions may occur or tumour shrinkage may occur. Furthermore, the strength of the various respiratory muscles can vary from day to day, as can the intra-abdominal pressure.

Currently, ART for lung carcinomas is carried out as part of patient care in the radiotherapy clinic at the University Hospital Essen. Patients are irradiated during repeated breath-holding manoeuvres in deep inspiration. The pure irradiation time takes about 1.5 minutes. The breath-holding manoeuvre is practised several times before the daily irradiation. An optical surface detection device is available for this purpose, which is used to compare the body surface in the patient's thorax area on the treatment table with the target surface to be achieved during radiotherapy planning, which took place days before the current fraction. If the target surface is reproducibly achieved, a conebeam CT is taken to determine the current tumour extent and the deformations occurring in comparison to the dose distribution to be applied. For this purpose, the normal tissues heart, lung and tracheal tree are automatically contoured by the Ethos therapy system in the cone-beam CT. A specialist physician and a physicist are present at the Ethos device during this process. These organ contours are used to determine the extent of the current target volume and the adaptive radiotherapy plan is adjusted to the new target volume. If the current tumour extent is not sufficiently covered by the initial radiotherapy plan planned for the series with its planned tolerances, or if the surrounding normal tissue is exposed to too much radiation, then the online adaptive radiotherapy plan for the current treatment is selected by the specialist. Otherwise, the initial radiotherapy plan is used by the planning CT as for IGRT.

The aim of this study is to treat 30 patients in ART readiness on the Ethos therapy device over 10 radiotherapy fractions. The dose distribution is always compared with the adaptive and the initial series plan on the anatomy of the day by the specialist and medical physics expert. The ART plan is then applied with dosimetric advantages. The aim of this study is to prospectively analyse in how many patients safety margins around the clinical target volume can be reduced with ART compared to IGRT. After the first 7 of the 10 fractions to be administered in ART readiness, the dose is accumulated over these fractions. The percentage of patients who benefit from ART will be determined prospectively. The criterion for a relevant benefit from ART is the effective uniform dose (EUD) in the target volume with the accumulated dose distribution across the 7 fractions. If the EUD is below 95% of the target dose with IGRT and above 95% of the target dose with ART, then an advantage is determined with ART. Such dose accumulations accompanying a radiotherapy series were not possible in the past. Patients with a benefit from ART receive ART for the further fractions of the series, while the others continue to be treated with IGRT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSCLC/SCLC ≥18 years of age in stage III or IV, oligometastatic, for whom the indication for neoadjuvant or definitive radiotherapy/radiotherapy/chemotherapy has been established in the certified lung tumour board.

Exclusion Criteria:

* Patients who are unable to perform a reproducible breath-hold manoeuvre on inspiration are not included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced non-small cell or small-cell lung cancer, respectively, to be treated with standard fractionation and dosage on the ETHOS therapy device after the indication (neoadjuvant/ definitive radiotherapy) has been determined in the multidisciplinary tumour board.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Advantage of ART over IGRT | 1.5 years
  In more than 50% of patients receiving definitive surgery-replacing or preoperative radiotherapy for locally advanced lung cancer, is it possible to reduce the planning margins around the clinical target volume (CTV) to compensate for movement and deformation with online-adaptive radiotherapy (ART) compared to IGRT?

SECONDARY OUTCOMES:
Determination of the percentage of patients who benefit from ART for lung cancer. | 1.5 years
  Exploratory analysis of factors that lead to an advantage of ART: Tumour shrinkage, variation in breath depth from day to day, localisation of the tumour in the lower lobe, previous lung disease, e.g. chronic obstructive pulmonary disease (COPD).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Stuschke, MD, Study Director — Klinik für Strahlentherapie, Universitätsklinikum Essen
Locations (1):
- Klinik für Strahlentherapie, Universitätsklinikum Essen, Essen, North Rhine-Westphalia, Germany